CLINICAL TRIAL: NCT01647789
Title: A Phase I/II, Multicenter, Open-label Dose Finding Study of Oral CFG920 in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Oral CFG920 in Patients With Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCFG920X2101; 2012-001961-33 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-24 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer, castration resistant,
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CFG920 (Experimental)
  Interventions: Drug: CFG920

INTERVENTIONS:
Drug: CFG920

SUMMARY:
This study was supposed to have assessed the safety and preliminary antitumor activity of CFG920, a new CYP17 inhibitor in castration resistant prostate cancer patients who are abiraterone naive or abiraterone resistant.

The study was terminated after Phase I (dose escalation phase) and Phase II part of the study was not initiated. Novartis voluntarily terminated this study and hence stopped further enrollment of patients into this study. As the decision to terminate the study was not due to any safety issues, the patients enrolled in the study by the time of this decision were allowed to continue with treatment per the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of castration resistant prostate cancer
* Documented metastases
* ECOG performance status 0 or 1
* Documented progression following the Prostate Cancer Working Group 2 guidelines
* Fresh or archived tumor sample

Exclusion Criteria:

* Impaired cardiac function
* Uncontrolled hypertension despire appropriate medical therapy
* History of pituitary or adrendal dysfunction
* Chronic steriod therapy other than daily use of 10mg prednisone
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral CFG920
* Brain metastases that have not been adequately treated
* Malignant disease other than that being treated in this study
* Laboratory abnormalities as specified in the protocol Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose limiting toxicities (DLT) | 28 days (from the time of first dose)
  Phase l; cycle = 28 days
Incidence rate of patients with Prostate Specific Antigen (PSA) response | >= 12 weeks
  Phase ll only

SECONDARY OUTCOMES:
Number of adverse events (AEs) | 18 months
  Phase l, Phase ll
PK parameters | 18 months
  Phase l, Phase ll
Prostate Specific Antigen (PSA) response (≥50% in PSA reduction) | 18 months
  Phase l only
Progression free survival (PFS) | baseline, until disease progression up to 6 months (6 cycle)
  Phase ll only; cycle = 28 days
Number of serious adverse events (SAEs) | 18 months
  Phase l, Phase ll
Time to PSA progression | up to 2 months (cycle 2)
  Phase ll; cycle = 28 days
Overall Response rate (ORR) | up to 2 months (cycle 2)
  Phase ll
Radiological Time to Progression (rTTP) | baseline, until date of documented disease progression
  Phase ll only
Prostate Specific Antigen (PSA) response (≥30% in the PSA reduction) | 18 months
  Phase ll only
Best PSA response at any time during the study | 18 months
  Phase ll only

OTHER OUTCOMES:
Evaluation of serum hormone levels | 18 months
  Phase I, Phase II
Correlate plasma exposure parameters of CFG920 and serum hormones | 18 months
  Phase I, Phase II
Evaluate moleculare profiles | 18 months
  Phase I, Phase II

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (4):
  - UCSF Medical Center Dept of Oncology, San Francisco, California
  - Cancer Therapy & Research Center UT Health Science Center InstituteForDrugDevelopment(2), San Antonio, Texas
  - Seattle Cancer Care Alliance Dept. of SCCA, Seattle, Washington
  - University of Wisconsin Univ Wisc, Madison, Wisconsin
- Novartis Investigative Site, Bouge, Belgium
- Novartis Investigative Site, Hamilton, Ontario, Canada
- Novartis Investigative Site, Barcelona, Catalonia, Spain